CLINICAL TRIAL: NCT07135128
Title: A Clinical Study of [225Ac]Ac-FAPI-XT(XT117) Injection in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xiaorong Sun (Other)
Responsible Party: Sponsor-Investigator, Xiaorong Sun, Director of Nuclear Medicine Department, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2024-366-01
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 225Ac-FAPI-XT treatment (Experimental)
  Interventions: Drug: 225Ac-FAPI-XT

INTERVENTIONS:
Drug: 225Ac-FAPI-XT — Patients will receive [225Ac]Ac-FAPI-XT(XT117) administration at an interval of 6 weeks between each dose.

SUMMARY:
This is a single-center, single-arm clinical study to evaluate the safety, tolerability and preliminary efficacy of [225Ac]Ac-FAPI-XT injection in patients with FAP-positive advanced solid tumors.

DETAILED DESCRIPTION:
A Clinical Study to Evaluate the Safety, Tolerability, Dosimetry and Preliminary Efficacy of [225Ac]Ac-FAPI-XT Injection in FAP-positive Patients With Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old Eastern Cooperative Oncology Group (ECOG) Performance status 0 to 1 Confirmed as malignant solid tumor by histopathology Have measurable lesions based on RECIST 1.1 Have failed standard treatment (disease progression or intolerance) or lack standard treatment Positive FAP expression confirmed by FAP PET/CT Sufficient bone marrow capacity and organ function

Exclusion Criteria:

* High intensity and large amounts of off-target uptake by FAP molecular imaging Previous systemic antitumor therapy (including prior chemotherapy, radiotherapy, immunotherapy, and other investigational drugs) ≤28 days before receiving study therapy; previous treatment with Chinese medicine with anti-tumor indications within 2 weeks before receiving study therapy Uncontrolled diabetes, with baseline fasting blood glucose > 2×ULN Clinically significant serious cardiovascular disease, including but not limited to: a. >Grade II congestive heart failure as per New York Heart Association (NYHA) ; b. Unstable angina pectoris or myocardial infarction within 6 months before the first administration of the study drug; c. Severe arrhythmia within 6 months prior to the first administration; d. Poorly controlled hypertension (patients who keep the blood pressure to ≤ Grade 2 hypertension [CTCAE5.0] with hypotensor are allowed for enrollment); e. QTc>450 ms (male) or 470 ms (female), congenital prolonged QT syndrome, and use of medications that prolong QT Clinically serious thromboembolic disease within 6 months prior to the first administration of the study drug Major surgery within 4 weeks prior to the initial administration of the study drug History of severe gastrointestinal ulcers or perforations or history of intestinal obstruction within 6 months prior to the first administration Active infection requiring systemic treatment (oral or intravenous administration) within 2 weeks prior to the first administration, except for topical treatment History of non-infectious interstitial lung disease (ILD), such as idiopathic pulmonary fibrosis, idiopathic interstitial pneumonia, pneumoconiosis, and drug-related interstitial pneumonia, or severe impairment of lung function Had other malignancies within 5 years prior to screening (except clinically cured early stage malignancies)

Primary central nervous system (CNS) tumor or symptomatic CNS metastasis, expect:

Subjects with asymptomatic brain metastases; Subjects whose CNS lesions were stable for ≥4 weeks after local treatment and who stopped glucocorticoid or anticonvulsant therapy at least 2 weeks prior to study drug administration could be enrolled; Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events | Through study completion, assessed up to 2 years
  adverse events Incidence and severity of treatment emergent adverse events will be assessed as per CTCAE v5.0.
Dose-limiting toxicity（DLT） | Through study completion, assessed up to 2 years
  Incidence and severity of dose-limiting toxicities.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Through study completion, assessed up to 2 years.
  Overall Response Rate (ORR) was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR). ORR was based on RECIST 1.1 response for patients with measurable disease at baseline.(based on RECIST 1.1).
Duration of Response (DOR) | Through study completion, assessed up to 2 years.
  Duration of Response (DOR) was defined as the duration between the date of first documented Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) and the date of first documented radiographic progression or death due to any cause .(based on RECIST 1.1).
Disease Control Rate (DCR) | Through study completion, assessed up to 2 years
  Disease control rate (DCR) was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) according to RECIST v1.1.
Progression Free Survival (PFS) | Through study completion, assessed up to 2 years.
  PFS is defined as the interval from the date of first dosing to the date of first demonstrated disease progression, or to the last date of known progression-free condition of the patient, or to the date of death (based on RECIST 1.1).

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Shandong First Medical University, Jinan, Shandong, China